CLINICAL TRIAL: NCT06441812
Title: A Multicenter, Single-group Phase II Clinical Study to Evaluate the Long-term Safety, Pharmacodynamics and Efficacy of Multiple Subcutaneous Injections of SHR-1703 in Eosinophilic Asthma Patients
Brief Title: A Study to Evaluate the Long-term Safety, Pharmacodynamics and Efficacy of SHR-1703 in Eosinophilic Asthma Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1703-202
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Eosinophilic Asthma Patients

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-1703 Injection (Experimental)
  Interventions: Drug: SHR-1703 Injection

INTERVENTIONS:
Drug: SHR-1703 Injection — SHR-1703 Injection

SUMMARY:
The purpose of this study is to evaluation the long-term Safety, Pharmacodynamics and Efficacy of SHR-1703 in Eosinophilic Asthma Patients

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age, Male or Femal.
2. A minimum weight of 40kg.
3. Subjects with the clinical features of asthma that meets the diagnostic criteria of the "Guidelines for the Prevention and Treatment of Bronchial Asthma (2020 Edition)" and has a medical history of at least 1 year.
4. Documentation of current asthma controller medication [medium or high dose ICS and at least one of additional controller such as long-acting muscarinic antagonist (LAMA), long-acting beta2-agonist (LABA) and leukotriene receptor antagonist (LTRA)] for at least 1 stable month before first administration of SHR-1703.
5. At least one confirmed history of exacerbation within one year of initial administration of SHR-1703, occurring during the use of medium and high daily dose ICS.
6. Absolute count of eosinophils must be ≥0.15×109/L at visit 0 and visit 1.
7. A pre-bronchodilator FEV1 <85% and ≥30% predicted at visit 0 and visit 1.
8. Female subjects with fertility agree to have no plan pregnancy and voluntarily adopt high-efficiency contraception measures from signing the informed consent form to 14 months after the last dose of SHR-1703, and male subjects with fertility as partners agree to have no plan pregnancy and voluntarily adopt high-efficiency contraception measures between the first dose of SHR-1703 and the last visit in the study.
9. Subjects must be able to give written informed consent prior to participation in the study.

Exclusion Criteria:

1. Presence of a clinically important lung condition. This includes but is not limited to current infection, bronchiectasis, pulmonary fibrosis or a history of lung cancer.
2. A known immunodeficiency.
3. Presence of a clinically significant and uncontrolled serious cardiovascular and cerebrovascular disease, including but not limited to myocardial infarction, unstable angina, heart failure, stroke, and subarachnoid haemorrhage.
4. Within the first 4 weeks before visit 0, presence of exacerbation of allergic rhinitis or sinusitis, or a history of infections with clinical significance and/or requiring clinical intervention, including but not limited to respiratory infections.
5. A known parasitic infection within the first 6 months before visit 0.
6. A malignancy history within the first 5 years before visit 0 (Subjects that had localized basal carcinoma of the skin or cervical carcinoma in situ which was resected for cure will not be excluded).
7. Blood donation or significant blood loss (≥ 400ml) within the first 4 weeks before visit 0, or infusion of blood products or immunoglobulins.
8. Use systemic immunosuppressants (excluding systemic glucocorticoids used for asthma treatment and for non asthma treatment for less than 3 days) or immunomodulators, or biologics or Th2 cytokine inhibitors, including but not limited to methotrexate, cyclosporine, interferon-α, anti IL-5 monoclonal antibodies (including SHR-1703), anti IL-4R monoclonal antibodies, anti TSLP monoclonal antibodies, anti IgE monoclonal antibodies, metformin, etc., and within 5 half-lives of the drug before the first administration (refer to the longer drug instructions; for those with unknown half-lives, 12 weeks before the first administration shall prevail);
9. Subjects who have previously participated in any study and received Investigational Product within the first 30 days before visit 0.
10. There was a surgical plan or other treatment measures that the researcher believed may affect the subject's evaluation during the study period.
11. Laboratory examination shows obvious abnormalities at visit 0 and visit 1:

    1. White blood cell count (WBC) <3.0×109/L;
    2. Hemoglobin≤90g/L；
    3. Platelet<100×109/L；
    4. Alanine aminotransferase (ALT)>2×ULN (upper limit of normal);
    5. Aspartate aminotransferase (AST) >2×ULN；
    6. Total bilirubin (TBIL)>1.5×ULN;
    7. Prothrombin time (PT) >ULN+3s；
    8. Creatinin>1.5×ULN;
    9. Active hepatitis B (positive for hepatitis B virus deoxyribonucleic acid (HBV DNA) in peripheral blood), or positive for hepatitis C virus antibody, or positive for human immunodeficiency virus (HIV) antibody, or positive for treponema pallidum antibody；
12. ECG QTc>450ms or other clinically significant abnormal results that may pose significant safety risks to the subjects at visit 0 or visit 1；
13. A history of drug addicts or substance abuse within 1 years prior to Visit 0；
14. Subjects who are pregnant (positive HCG test at visit 0 or visit 1) or breastfeeding should not be enrolled if they plan to become pregnant during the time of study participation；
15. Subjects with a known allergy or intolerance to anti IL-5 monoclonal antibody or other biologic；
16. Other reasons determined by the researcher as unsuitable for participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-07-19 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Adverse Events in main peroid，about 1 year | about 1 year

SECONDARY OUTCOMES:
Absolute count of eosinophils , about 1 year | about 1 year
Change of FEV1 、FEV1%pred、FVC、PEF，about 1 year. | about 1 year.
Change of Fractional Exhaled Nitric Oxide (FeNO) ，about 1 year. | about 1 year.
Questionnaire about asthma，about 1 year . | about 1 year .
Frequency and time of asthma exacerbation , about 2 years | about 2 years
Reduction in asthma controller , about 1 year | about 1 year
Asthma remission, about 2 years | about 2 years
Daily OCS use and reduction, about 1 year. | about 1 year.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided